CLINICAL TRIAL: NCT06952959
Title: Using Professional Intelligent Skin Analyzers to Analyze the Effects of Cosmetic Acupuncture on Skin Health and Aging: A Randomized Controlled Trial
Brief Title: The Effects of Cosmetic Acupuncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chia-Hui Lin, Attending Physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC2-018
Record Dates: First submitted 2025-04-10; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aging; Skin Health
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cosmetic acupuncture group (Experimental): accept treatment session
  Interventions: Other: Acupuncture
- Waitinglist for cosmetic acupuncture group (Other): wait for 3 weeks then accept the same treatment session
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Cosmetic acupuncture

SUMMARY:
The study recruited 40 subjects and divided them into an intervention group and a waiting list group in a 1:1 ratio using a randomized controlled trial. The changes in skin health and aging-related indicators before and after TCM cosmetic acupuncture treatment were analyzed. The subjects are of all genders and aged between 30 and 60 years old. The TCM cosmetic acupuncture treatment is arranged twice a week for a three-week course. The study will conduct a skin test before and after the TCM cosmetic acupuncture, and use the Antera 3D smart skin detector to comprehensively evaluate the subjects' skin condition. Antera 3D Skin Detector can detect multiple skin indicators, including wrinkle depth, skin tone uniformity and subtle changes in the skin surface, melanin, red pigment, etc. After the treatment, the subjects' acceptance and satisfaction with TCM cosmetic acupuncture were collected.

ELIGIBILITY:
Inclusion Criteria:

* both female and male
* 30 to 60 years old
* never had acupuncture beauty treatment, or the last time they had acupuncture beauty treatment has been more than six months.

Exclusion Criteria:

* medical cosmetic fillers on their face
* cosmetic surgery
* needle sickness
* afraid of acupuncture
* wounds on the facial skin
* poor wound healing
* abnormal coagulation function
* severe diabetes
* keloids
* dialysis
* cancer patients undergoing chemotherapy or radiotherapy
* pregnant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Face Skin Texture | Intervention group: the 1st, 4th week; waiting list group: the 1st, 4th, and 7th week.
  Professional Intelligent Skin Analyzers accurately locate the comparison before and after cosmetic acupuncture sessions, showing high accuracy and reproducibility, analyzing Ra value (unit: µm) as arithmetic mean roughness of the skin's contours.
Face Skin Color | Intervention group: the 1st, 4th week; waiting list group: the 1st, 4th, and 7th week.
  Professional Intelligent Skin Analyzers accurately locate the comparison before and after cosmetic acupuncture sessions, showing high accuracy and reproducibility, analyzing L*a*b value (no unit) as the skin's color. (L*: Lightness, a*: Red/Green Value, b*: Blue/Yellow Value)
Face Pore Size | Intervention group: the 1st, 4th week; waiting list group: the 1st, 4th, and 7th week.
  Professional Intelligent Skin Analyzers accurately locate the comparison before and after cosmetic acupuncture sessions, showing high accuracy and reproducibility, analyzing average pore volume (unit: mm²).

SECONDARY OUTCOMES:
The Questionnaire of satisfaction and acceptance of cosmetic acupuncture | Intervention group: the 4th week; waiting list group: the 7th week.
  The questionnaire include three domains: 1. Visual Analogue Scale score measures pain intensity. The VAS consists of 10 points, with two end points representing 0 ("no pain") and 10 ("pain as bad as it could possibly be"). 2. The acceptance of cosmetic acupuncture has 0~4 points, 0 representing "unacceptable" and 4 representing "totally acceptable". 3. Facial Check Sheet(FCS) has 12 items about the satisfaction of the improvement of face appearance including wrinkles, laxity, facial shape, and pigmented spots, and so on. 0 representing "very dissatisfied" and 4 representing "very satisfied". Subjects can also choose "no need to pay attention" if they don't have the concerned problems of appearance.

CONTACTS AND LOCATIONS:
Locations (1):
- China medical university hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No